CLINICAL TRIAL: NCT03185988
Title: Multicenter, Phase II Study of Chemotherapy in Combination With Trastuzumab in Patients of Pretreated, HER2 Positive, Relapse or Metastatic Carcinoma of Digestive System
Brief Title: Anti-HER2 Therapy in Patients of HER2 Positive Metastatic Carcinoma of Digestive System
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shen Lin (Other)
Responsible Party: Sponsor-Investigator, Shen Lin, Prof., Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG2006
Record Dates: First submitted 2017-05-16; First posted 2017-06-14 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Targeted Therapy; HER2; Biliary Tract Cancer; Esophageal Squamous Cell Carcinoma; Colorectal Cancer
Keywords: Human epidermal growth factor receptor 2; Biliary tract cancer; Esophageal squamous cell carcinoma; Targeted therapy; colorectal cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Esophageal Squamous Cell Carcinoma; Colorectal Neoplasms | interventions — Drug Therapy; Trastuzumab; 26S proteasome non-ATPase regulatory subunit 13; JPT1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GI tumor beyond CRC, ESCC, BTC,GC&GEJA (Experimental): HER2 positive GI tumor beyond CRC, ESCC, BTC,GC&GEJA
  Interventions: Drug: chemotherapy in combination with trastuzumab for arm1
- Esophageal squamous cell carcinoma (Experimental): HER2 positive Esophageal squamous cell carcinoma
  Interventions: Drug: chemotherapy in combination with trastuzumab for arm2
- Biliary tract cancer (Experimental): HER2 positive Biliary tract cancer
  Interventions: Drug: chemotherapy in combination with trastuzumab for arm3
- Colorectal cancer (Experimental): HER2 positive and RAS/BRAF wild type colorectal cancer
  Interventions: Drug: chemotherapy in combination with trastuzumab for arm4

INTERVENTIONS:
Drug: chemotherapy in combination with trastuzumab for arm1 — Arm1: GI tumor beyond CRC, ESCC, BTC and GC&GEJA Trastuzumab (Herceptin ®): 6 mg/kg every 3 weeks (8 mg/kg as loading dose at 1st administration), iv, d1.The first infusion is to be given over 90 minutes, and subsequent infusions are to be given over 30 minutes if the first infusion is well tolerated.Combined chemotherapy (by investigator's choice)
  Arms: GI tumor beyond CRC, ESCC, BTC,GC&GEJA
Drug: chemotherapy in combination with trastuzumab for arm2 — Arm2: esophageal squamous cell carcinoma (ESCC) Trastuzumab (Herceptin ®): the same as above Combined with Irinotecan: 120 mg/m2 IV, day 1 and day 8, every 3 weeks.
  Arms: Esophageal squamous cell carcinoma
Drug: chemotherapy in combination with trastuzumab for arm3 — Arm 3: biliary tract cancer (BTC) Trastuzumab (Herceptin®): the same as above Combined chemotherapy (by investigator's choice) The combined chemotherapy of cohort 1 and 3 is Irinotecan: 120 mg/m2 IV, day 1and day 8, every 3 weeks.
  OR 5-Fu: 720 mg/m2/day, continuous IV. Infusion over 5 days, every 3 weeks. OR Capecitabine(Xeloda®):1000 mg/m2 bid, d1-d14, every 3 weeks. The chemotherapy regimen is chosen at the Investigator's discretion and can be determined on an individual patient basis. Special cases should be discussed with the principal investigator.
  Arms: Biliary tract cancer
Drug: chemotherapy in combination with trastuzumab for arm4 — Trastuzumab (Herceptin ®): same as above Combined with Irinotecan: 120 mg/m2 iv, day 1and day 8, every 3 weeks. OR Capecitabine(Xeloda®)1000 mg/m2 bid, d1-d14, every 3 weeks. OR Irinotecan: 120 mg/m2 iv, day 1and day 8 and Capecitabine(Xeloda®)1000 mg/m2 bid, d1-d14, every 3 weeks (by investigator's choice)
  Arms: Colorectal cancer

SUMMARY:
To seek the efficacy signals of trastuzumab in combination with chemotherapy in pretreated patients of HER2 positive, relapse or metastatic carcinoma of digestive system as response rate (RR) determined by the Investigator using RECIST 1.1, and provide evidence for phase III clinical trial.

DETAILED DESCRIPTION:
Human epidermal growth factor receptor 2, (HER2) is overexpressed /amplified in multiple carcinomas, for example, gastric cancer(GC), gastroesophageal junction adenocarcinoma(GEJA),and breast cancer.And HER2 is closely related to tumor proliferation &metastases.About 90% Chinese esophagus cancer are squamous cell origin. The reported HER2 overexpression ranged from 5-30%, Beijing cancer hospital reported an 11% positive rate. The variety of HER2 positive rate may because of the absence of standard HER2 testing criteria. The current treatment for metastatic Esophageal squamous Cell Carcinoma (ESCC) is not satisfactory. Fluorouracil and platinum are considered as first line standard of care (SOC) with a 20-30% RR and 7-9 months overall survival (OS). In second line setting, there is no SOC in china. And the efficacy is not satisfactory. Esophageal adenocarcinoma has a higher HER2 positive rate of 14%, but no data reported of using trastuzumab in these patients in China. Biliary tract cancer (BTC), including intrahepatic/extrahepatic cholangiocarcinoma and Gallbladder cancer (GBC) is very aggressive, total 5y survival is less than 5% for unresectable patients. GBC is account for approximately 2/3 of BTC, and it's estimated the incidence in china is 52800 and the mortality is 40700 in 2015. Most patients are diagnosed in advanced stage and lose the opportunity of surgery. However, there is no SOC for unresectable BTC, gemcitabine plus platinum provided a 30% RR and 10 month OS. In second line treatment, no differences were seen between various experimental agents. The reported HER2 positive rate range from 5.1% to 57% in biliary duct cancer and 4.7% to 64% in GBC. Researchers reported her2 amplification is related to tumor stage and lymph nodes metastasis in 221 BTC patients. Another study reported a 16.6% positive rate and worse prognosis with a sample size of 230 GBC patients. Meanwhile, HER2 pathway mutation rate reached 37%. All imply that BTC may be the potential anti HER therapy population. Besides, other digestive system tumor has low HER2 positive rate (Small intestinal cancer 0.9-3%; hepatocellular carcinoma 2.4%; Pancreatic cancer 3%; etc.). However, the patient pool is large and has no SOC in second Line. Whether these HER2 + patients can gain benefit form anti- her treatment is worth investigating. In 2016 American Society of Clinical Oncology (ASCO), a study reported that using trastuzumab and pertuzumab combination, 35% metastatic colorectal cancer (CRC) and 50% BTC patients who heavily pretreated had objective response. However, china doesn't have studies for these patients. .

The concurrent basket trial will explore the efficacy and safety of trastuzumab with chemotherapy in Chinese patients of pretreated, HER2 positive, relapse or metastatic carcinoma of digestive system.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Male and female patients aged from 18 to 75 years
* Histologically confirmed Colorectal cancer,Esophagus squamous cell carcinoma, biliary tract cancer, and digestive system tumor beyond CRC and GC&GEJA with the following specifications:

  * genetic testing conformed KRAS/NRAS/BRAF all wild type for colorectal cancer
  * Detection of a carcinoma with HER2 3+ (IHC) or HER2 2+ (IHC) with amplification proven by fluorescence in situ hybridization(FISH), silver in situ hybridization（SISH） or chromogenic in situ hybridization（CISH） using gastric cancer criteria by an accredited local pathologist.
  * Relapse or metastatic diseases, at least one measurable lesion according to RECIST 1.1, anticipated survival ≥ 12 weeks.
  * ECOG Performance status 0-1.
  * Patients who failed at least first line systemic therapy.
  * Adequate organ function as determined by the following laboratory results:
  * Absolute neutrophil count ≥1500 cells/mm3,
  * Platelet count ≥ 90,000 cells/mm3,
  * Hemoglobin ≥9.0 g/dL
  * Total bilirubin ≤ 1.5 upper limit of normal (ULN).
  * serum glutamate oxaloacetate transaminase(SGOT,AST), serum glutamate pyruvate transaminase(SGPT,ALT) < 2.5 ULN without liver metastases; < 5 ULN with liver metastases.
  * serum creatinine < 1.5
  * ULN OR creatinine clearance ≥ 40 mL/ min.
* If able to reproduce, patients must be willing to use highly effective methods of contraception during treatment and for 7 months after the end of treatment.

Exclusion Criteria:

* Known hypersensitivity against treatment regimen.
* Baseline left ventricular ejection fraction(LVEF) < 50% (measured by echocardiography or MUGA).
* Previous anti-her treatment.
* Immune therapy, biological therapy or any participation in clinical trial in previous two weeks.
* Surgery and not recovered in previous three weeks
* Clinical evidence of brain metastases, or uncontrolled epilepsy.
* Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
* Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, New York Heart Association(NYHA) III-IV; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; unstable angina pectoris, myocardial infarction or high risk uncontrollable arrhythmias.
* Long term or high dose corticosteroids administration ( inhalation or short term oral administration for antiemesis and orexigenic is allowed)
* Patients of legally incapacity or of medical and ethical reasons not fit for study.
* Pregnant or lactating, or intending to become pregnant during the study.
* Jaundice, ascites, and / or alkaline phosphatase ≥3 × ULN; and / or ≥3 grade (CTC-AE) of persistent proteinuria, urinary protein / creatinine ratio> 3.5g / 24 hours or renal failure need blood or peritoneal dialysis.
* Presence of > grade 2(CTC-AE) persistent infection; unhealed wounds, ulcer or fracture, or patients with a history of organ transplant.
* Evidence of coagulation disorders. Like presence ≥grade 3 (CTC-AE) bleeding events.
* Known HIV or hepatitis B virus(HBV), hepatitis C virus(HCV) infection.
* Any > grade 1 unresolved toxicity due to previous treatment (CTC-AE), except for alopecia, anemia and hypothyroidism).
* Not suitable for the study evaluated by investigators
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* History of exposure to the following cumulative doses of anthracyclines:

  * Doxorubicin > 500 mg/m2 OR Epirubicin > 720 mg/m2.

    * If another anthracycline or more than one anthracycline has been used, then the cumulative dose must not exceed the equivalent of 500 mg/m2 doxorubicin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Response Rate(RR) for each cohort in intent to treat (ITT) population | baseline up to death or disease progression,which ever occurs first(up to approximately 8.5 years)
  The percentage of patients, whose tumor volume in first time shrink to pre-defined criteria, including CR and PR

SECONDARY OUTCOMES:
Disease control rate | baseline up to death or disease progression,which ever occurs first(up to approximately 8.5 years)
  The percentage of patients who achieve complete remission(CR) or partial remission (PR) or stable disease(SD) determined by the RECIST v1.1 criteria.
best overall response | 10-30 weeks
  The percentage of patients who achieve either a CR or PR as determined by the RECIST v1.1 criteria based on investigator's assessment that is confirmed by a repeat assessment performed no less than 4 weeks after the criteria for response are first met.
Progression free survival | baseline up to death or disease progression,which ever occurs first(up to approximately 8.5 years)
  Defined as the initiation of treatment to the day of first documentation of PD or date of death, whichever occurs first.
Overall survival | baseline up to death or disease progression,which ever occurs first(up to approximately 8.5 years)
  Is the time from the initiation of treatment to the date of death from any cause.
time to response | 6-30 weeks
  Defined as the initiation of treatment to the day of first documentation of response.
  Only patients who achieve an objective response will be included in the analysis.
duration of response | 6-30 weeks
  Defined as the time from the date of the first documented objective response to the date of first documented PD or death, whichever occurs first. Only patients who achieve an objective response will be included in the analysis.
time to progression(TTP) | 6-30 weeks
  Defined as the initiation of treatment to the day of first documentation of PD.
Quality of Life by Eastern Cooperative Oncology Group(ECOG)performance status( PS) scoring criteria | Day 1 of each 21-day treatment cycle up to 28 days and 60-90 days after Day 1 of last treatment cycle(up to approximately 8.5 years)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | baseline up to approximately 8.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Master, Principal Investigator — Director
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu T, Wang X, Xin Y, Wang Z, Gong J, Zhang X, Li Y, Ji C, Sun Y, Zhao F, Huang D, Bai Y, Li J, Shen L. Trastuzumab Combined with Irinotecan in Patients with HER2-Positive Metastatic Colorectal Cancer: A Phase II Single-Arm Study and Exploratory Biomarker Analysis. Cancer Res Treat. 2023 Apr;55(2):626-635. doi: 10.4143/crt.2022.1058. Epub 2022 Dec 23. PMID 36550683